CLINICAL TRIAL: NCT03610139
Title: Longitudinal Effect of Vitamin D3 Replacement on Cognitive Performance and MRI Markers in Multiple Sclerosis Patients: A Single-Blind Randomized Clinical Trial
Brief Title: Longitudinal Effect of Vitamin D3 Replacement on Cognitive Performance and MRI Markers in Multiple Sclerosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Hala Darwish, Associate Professor - Hariri School of Nursing / Managing Director - Abu-Haidar Neuroscience Institute / Managing Director - Nehme and Therese Tohme Multiple Sclerosis Center, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BIO-2017-0395
Record Dates: First submitted 2018-07-13; First posted 2018-08-01 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Clinically Isolated Syndrome; Clinically Isolated Syndrome, CNS Demyelinating; Vitamin D3 Deficiency
Keywords: cognitive performance; vitamin D3 replacement; Lebanon
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Demyelinating Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: One of the co-investigators who will perform the MRI segmentation and analysis will be blind to the participants' treatment allocation.
  Research assistants who will administer the cognitive tests to all participants will be blind to the participants' treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low dose vitamin D3 supplementation (Active Comparator): Patients in this group will take 800 IU daily dose of vitamin D supplementation. They will be kept on 800 IU for 6 months. If they still had low vitamin D at 3 months, they will be asked about their adherence to the supplement, the investigators will remind them to take it as prescribed, and the investigators will keep the 800 IU vitamin D supplement dose for another 3 months. If they were still deficient at 6 months, the investigators will switch them to 10,000 IU weekly dose.
  Interventions: Dietary Supplement: Vitamin D3
- high dose vitamin D3 supplementation (Experimental): Patients in this group will take 50,000 IU weekly dose of vitamin D supplementation. Patients who will reach normal serum vitamin D level, between 40-80 ng/ml, at 3 or 6 months will be asked to decrease their Vitamin D3 supplementation as follows: Those who will reach levels between 40-60ng/ml will be switched to 10,000 IU three times per week, and those who reach levels between 60-80 ng/ml will be switched to 10,000 IU once weekly.
  If they did not have any improvement in their levels of vitamin D at 3 or 6 months, they will be asked about their adherence to the supplement and the investigators will remind them to take it as prescribed and the investigators will keep them at the 50,000 IU weekly dose.
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — At baseline, patients with deficient 25(OH)D levels will be randomly assigned 1:1 to receive either the high dose or standard dose vitamin D supplementation.

SUMMARY:
This is a longitudinal single blind randomized trial to test the effects of high compared to low dose vitamin D3 supplementation on cognitive performance at 6 and 12 months, and MRI measures of 12 months duration. A cognitive assessment battery will be administered at baseline, 6 and 12 months. Related clinical data and information on depression and anxiety, lifestyle, and food sources of vitamin D and sun exposure among other variables will also be collected.

DETAILED DESCRIPTION:
Background: Multiple Sclerosis is strongly associated with low serum 25 hydroxy-vitamin-D (25(OH)D) and impaired cognitive performance. In our previous research, participants with low serum 25OHD levels showed significant improvements in visuo-spatial memory delayed recall after 3 months of vitamin D3 supplementation. In addition, serum 25(OH)D was significantly associated with this memory function at baseline and at 3 months. Therefore, the aim of this proposed study is 1) to evaluate the long-term effects 6 and 12 months of high (50,000 IU weekly then 10,000 IU weekly) compared to low dose (800 IU daily) vitamin D3 replacement on cognitive function in MS, and 2) to correlate it with the MRI brain measurements of the hippocampus and the frontal cortex volumes, as well as brain parenchymal fraction, and cerebellum. The investigators will then explore these MRI measures in MS patients with deficient 25(OH)D levels at baseline and at 12 months, and correlate it with their cognitive performance.

Methods: This is a longitudinal single blind randomized trial to test the effects of high compared to low dose vitamin D3 supplementation on cognitive performance at 6 and 12 months, and MRI measures of 12 months duration. A cognitive assessment battery, comprised of the Montreal Cognitive Assessment (only at baseline), Stroop, Symbol Digit Modalities Test, Brief Visual Memory Test, and Verbal Memory Test in Arabic, will be administered at baseline, 6 and 12 months. Related clinical data and information on depression and anxiety, lifestyle, and food sources of vitamin D and sun exposure among other variables will also be collected.

Expected results: MS patients with serum 25(OH)D deficiency who receive high dose vitamin D3 supplementation will demonstrate decreased cognitive impairment at 6 and 12 months post supplementation when compared to those who received low vitamin D3 dose and to their pre-supplementation status. The MRI findings are expected to be associated with cognitive performance at baseline, and serum 25(OH)D levels at baseline, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Males/ Females
* Age ≥ 18 years old
* Have a definite diagnosis of RRMS as per the revised McDonald 2010 or CIS.
* Untreated or on any MS therapy
* Showed no clinical evidence of relapses during the past month and disease duration not greater than 10 years.
* Subjects who have a serum vitamin D level below 25 ng/ml

Exclusion Criteria:

* All subjects using drugs associated with hypercalcemia.
* Pregnant and with history of primary hyper PTH.
* Subjects with hypercalcemia, renal dysfunction, malignancy, or granulomatous disease, dementia, traumatic brain injury, diagnosis of epilepsy or history of seizure, psychiatric disease other than anxiety and depression, or are found to be suicidal on screening, or taking psychoactive medications other than antidepressants
* Subjects who have a serum vitamin D level above 25 ng/ml
* Subjects who have not done an MRI scan up to 3 months before or after the baseline visit.
* Subjects who have a history of kidney stones
* Subjects with malabsorption
* Individuals with history of alcohol abuse/dependence and/or substance use/abuse/dependence will also be excluded from the study. Men who consume more than 15 drinks per week and women who consume more than eight drinks per week will be considered excessive alcohol consumers and will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Brief Visuospatial Memory Test-Revised (BVMT-R) scores at 6 months | 6 months
  It is a visuospatial memory test that is comprised of three memory trials (10 seconds each) followed by delayed recall trial after 25 minutes. It has been widely used as a quick measure of memory at bedside and in MS patients. The minimum score on each trial is 0 and the maximum score on each trial is 12. Higher values represent a better outcome.
Change from Baseline Arabic Verbal Memory Test (VMAT) scores at 6 months | 6 months
  It is a verbal memory test. It consists of 45 words that are distributed among 3 lists (List A, List B, and a Recognition List). Lists A and B are each composed of 15 words belonging to 3 semantic categories: vegetables, animals, and stationary. The recognition list is composed 45 words that include homonyms, shared or related words and unrelated words with respect to the previous two lists. The VMAT is administered as follows: List A Immediate Free Recall (5 trials) - List B Immediate Free Recall Trial - List A Short Delay Free Recall Trial - List A Short Delay Cued Recall Trial - List A Long Delay Free Recall Trial - List A Long Delay Cued Recall Trial. After 25 minutes of the last trial, List A Delayed Recognition Trial is administered. For each trial, the minimum total score is 0 and the maximum total score is 15. Higher scores represent a better outcome. For each trial except the recognition trial, repeated and intrusive words are counted separately.
Change from Baseline Symbol Digit Modalities Test (SDMT) scores at 6 months | 6 months
  It is a known and widely used speed of processing test. Oral SDMT will be administered; it does not require translation and has been used in Lebanon before. It consists of one trial. The minimum total score is 0 and the maximum total score is 110. Higher scores represent a better outcome.
Change from Baseline Stroop test scores at 6 months | 6 months
  It is a highly established test of attention. Subject is given a list of colors in black ink to read (Stroop 1), then a list of colors in their corresponding ink color (Stroop 2), and then finally a list of colors with incongruent ink colors (Stroop 3), the participant is expected to read the word without being affected by interfering mismatching color. The number of words read in a minute (minus the errors) is the dependent measure and interference will be calculated using the following equation: Interference = Stroop 3 - [(Stroop 1+Stroop 2)/2]. For each of the 3 lists, the minimum total score is 0 and the maximum total score is 100. Higher scores represent a better outcome. For the interference, the minimum score is -100 and the maximum score is 0. Higher scores represent a better outcome.
Change from Baseline Brief Visuospatial Memory Test-Revised (BVMT-R) scores at 12 months | 12 months
  It is a visuospatial memory test that is comprised of three memory trials (10 seconds each) followed by delayed recall trial after 25 minutes. It has been widely used as a quick measure of memory at bedside and in MS patients. The minimum score on each trial is 0 and the maximum score on each trial is 12. Higher values represent a better outcome.
Change from Baseline Arabic Verbal Memory Test (VMAT) scores at 12 months | 12 months
  It is a verbal memory test. It consists of 45 words that are distributed among 3 lists (List A, List B, and a Recognition List). Lists A and B are each composed of 15 words belonging to 3 semantic categories: vegetables, animals, and stationary. The recognition list is composed 45 words that include homonyms, shared or related words and unrelated words with respect to the previous two lists. The VMAT is administered as follows: List A Immediate Free Recall (5 trials) - List B Immediate Free Recall Trial - List A Short Delay Free Recall Trial - List A Short Delay Cued Recall Trial - List A Long Delay Free Recall Trial - List A Long Delay Cued Recall Trial. After 25 minutes of the last trial, List A Delayed Recognition Trial is administered. For each trial, the minimum total score is 0 and the maximum total score is 15. Higher scores represent a better outcome. For each trial except the recognition trial, repeated and intrusive words are counted separately.
Change from Baseline Symbol Digit Modalities Test (SDMT) scores at 12 months | 12 months
  It is a known and widely used speed of processing test. Oral SDMT will be administered; it does not require translation and has been used in Lebanon before. It consists of one trial. The minimum total score is 0 and the maximum total score is 110. Higher scores represent a better outcome.
Change from Baseline Stroop test scores at 12 months | 12 months
  It is a highly established test of attention. Subject is given a list of colors in black ink to read (Stroop 1), then a list of colors in their corresponding ink color (Stroop 2), and then finally a list of colors with incongruent ink colors (Stroop 3), the participant is expected to read the word without being affected by interfering mismatching color. The number of words read in a minute (minus the errors) is the dependent measure and interference will be calculated using the following equation: Interference = Stroop 3 - [(Stroop 1+Stroop 2)/2]. For each of the 3 lists, the minimum total score is 0 and the maximum total score is 100. Higher scores represent a better outcome. For the interference, the minimum score is -100 and the maximum score is 0. Higher scores represent a better outcome.

SECONDARY OUTCOMES:
Change from Baseline Magnetic Resonance Imaging Brain Markers of the Hippocampus volume at 12 months | 12 months
  Changes in baseline MRI brain measurements of the hippocampus volume will be assessed at 12 months.
Change from Baseline Magnetic Resonance Imaging Brain Markers of the frontal cortex volume at 12 months | 12 months
  Changes in baseline MRI brain measurements of the frontal cortex volumes will be assessed 12 months.
Change from Baseline Magnetic Resonance Imaging Brain Markers of the brain parenchymal fraction at 12 months | 12 months
  Changes in baseline MRI brain measurements of the brain parenchymal fraction will be assessed at 12 months.
Change from Baseline Magnetic Resonance Imaging Brain Markers of the Cerebellum at 12 months | 12 months
  Changes in baseline MRI brain measurements of the cerebellum will be assessed at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Darwish, PhD, RN, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- Nehme & Therese Tohme Multiple Sclerosis Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darwish H, Haddad R, Osman S, Ghassan S, Yamout B, Tamim H, Khoury S. Effect of Vitamin D Replacement on Cognition in Multiple Sclerosis Patients. Sci Rep. 2017 Apr 4;7:45926. doi: 10.1038/srep45926. PMID 28374837
- [Background] Balion C, Griffith LE, Strifler L, Henderson M, Patterson C, Heckman G, Llewellyn DJ, Raina P. Vitamin D, cognition, and dementia: a systematic review and meta-analysis. Neurology. 2012 Sep 25;79(13):1397-405. doi: 10.1212/WNL.0b013e31826c197f. PMID 23008220
- [Background] Darwish H, Zeinoun P, Ghusn H, Khoury B, Tamim H, Khoury SJ. Serum 25-hydroxyvitamin D predicts cognitive performance in adults. Neuropsychiatr Dis Treat. 2015 Aug 25;11:2217-23. doi: 10.2147/NDT.S87014. eCollection 2015. PMID 26346368
- [Background] van der Schaft J, Koek HL, Dijkstra E, Verhaar HJ, van der Schouw YT, Emmelot-Vonk MH. The association between vitamin D and cognition: a systematic review. Ageing Res Rev. 2013 Sep;12(4):1013-23. doi: 10.1016/j.arr.2013.05.004. Epub 2013 May 29. PMID 23727408